CLINICAL TRIAL: NCT06246032
Title: Impact of Modified Feeding Protocol on Neonatal Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Hanan AlQahtani, Clinical Dietitian, Imam Abdulrahman Bin Faisal University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-PGS-2023-03-443
Record Dates: First submitted 2024-01-05; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Preterm; Birth Weight; Feeding Disorder Neonatal
Keywords: Feeding protocol; Neonates; Preterm; Very low birthweight; NICU
MeSH Terms: conditions — Premature Birth; Birth Weight

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified feeding Protocol (Experimental): Prospective
  Interventions: Other: Modified feeding Protocol
- Current feeding Protocol (No Intervention): Retrospective data will be collected from medical record of patients undergo the current feeding protocol as follow
  Initiation of feeding (average):
  8.7cc/kg (6-12cc/kg)
  Advancement based on birthweight (average):
  <750g: 20cc/kg/d (17-24cc/kg/d) 750-999g: 29cc/kg/d (25-34cc/kg/d) 1000-1249g: 22cc/kg/d (20-24cc/kg/d) 1250-1499g: 24cc/kg/d (21-25cc/kg/d) 1500-1749g: 20cc/kg/d (18-21cc/kg/d) 1750-2000g: 34cc/kg/d (32-36cc/kg/d)
  Starting Human milk fortification when feed reach at 120cc/kg/d

INTERVENTIONS:
Other: Modified feeding Protocol — Initiation of feeding (fixed): 10cc/kg
  Advancement based on birthweight (fixed):
  <750g: 15cc/kg/d 750-999g: 20cc/kg/d 1000-1249g: 25cc/kg/d 1250-1499g: 25cc/kg/d 1500-1749g: 35cc/kg/d 1750-2000g: 35cc/kg/d
  Starting Human milk fortification when feed reach at 70cc/kg/d
  Arms: Modified feeding Protocol

SUMMARY:
The goal of this clinical trial is to compare modified feeding protocol and current feeding protocol on neonatal outcomes in preterm infants who born with weight less than 2kg.

The main questions it aims to answer are:

* Is Modified feeding protocol will decrease the duration of parenteral nutrition and length of hospital stay?
* Is Modified feeding protocol feasible, efficient, and safe in preterm infants?

Participants will undergo the modified feeding protocol since birth until discharge.

DETAILED DESCRIPTION:
two group in this study Prospective group: intervention group will undergo the modified feeding protocol Retrospective group: intervention group will undergo the current feeding protocol

Both group will have care as routine care to this kind of patients But the differ will be in feeding protocol as initiation rate, advancement rate, human milk fortification rate

The outcomes of both group will be compeered to meet the study objectives

ELIGIBILITY:
Inclusion Criteria:

* Birth weight (<2000g)
* Gestational Age (<37 week)

Exclusion Criteria:

* Metabolic Disorders
* Congenital Heart Diseases
* Chronic Lung Disease
* Congenital Anomalies (can related to feeding)
* Moderate to severe GERD
* Necrotizing enterocolitis stage 3 (surgical)
* Gastrointestinal surgery

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Length of Stay (LOS) | Up to 8 weeks
  Number of days that participant stayed at hospital
Duration of Total Parenteral Nutrition (TPN) | up to 2 weeks
  Number of days that participant received Total Parenteral Nutrition (TPN)

SECONDARY OUTCOMES:
Incidence of Necrotizing Enterocolitis | Up to 8 weeks
  Stage 2, Stage 3
Incidence of Feeding intolerance | Up to 8 weeks
  abdominal grith more than 2 cm, gastric residual 50% of the last feed.

CONTACTS AND LOCATIONS:
Overall Officials: Hanan AlQahtani, Master, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- Maternity and Children Hospital, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No